CLINICAL TRIAL: NCT07263620
Title: A Single-center, Exploratory Study on Predicting Neoadjuvant Therapy Efficacy and Prognosis in Pan-gastrointestinal Cancer Patients Based on Intratumoral Microbiome Characteristics and Their Functional Targets.
Brief Title: An Exploratory Study on Microbial Biomarkers Associated With the Efficacy of Neoadjuvant Therapy
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc20253994
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Digestive System Malignancies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pancreatic cancer
  Interventions: Other: This study is observational and involves no interventions.
- gastric cancer
  Interventions: Other: This study is observational and involves no interventions.
- colorectal cancer
  Interventions: Other: This study is observational and involves no interventions.

INTERVENTIONS:
Other: This study is observational and involves no interventions. — This study is observational and involves no interventions.

SUMMARY:
Digestive system malignancies are among the most common types of cancers in China, primarily including esophageal cancer, gastric cancer, pancreatic cancer, liver cancer, and colorectal cancer. According to the 2024 National Cancer Registry data released by the National Cancer Center of China (covering a population of 523 million), digestive system tumors (including colorectal, liver, gastric, and esophageal cancers) account for 28.49% of all new cancer cases and 31.77% of total cancer-related deaths in the country. Among these, the incidence and mortality burdens of gastric, esophageal, and liver cancers are significantly higher than the global average. Most patients are diagnosed at an advanced stage, with a five-year survival rate below 30%. This highlights that digestive system malignancies represent a major public health challenge in China, necessitating in-depth studies on their pathogenesis and the development of novel prevention and treatment strategies.

At present, radical surgical resection remains the only potentially curative option for digestive system cancers. However, for patients with locally advanced or late-stage disease, surgery alone yields limited efficacy. In recent years, chemotherapy-based neoadjuvant therapy has been increasingly applied in clinical practice to improve R0 resection rates and overall survival [4-6]. Nevertheless, current studies show that the response rate to neoadjuvant therapy remains modest, and there is a lack of precise strategies for identifying therapy-sensitive patient subgroups, resulting in a limited proportion of patients who truly benefit.

The gut microbiota, as an essential component of the human microecosystem, plays a critical role in tumor initiation, progression, metastasis, and therapeutic response. Given the anatomic location of digestive system cancers, the gut microbiota-being a major source of intratumoral microorganisms-interacts closely with the tumor microenvironment. Studies have revealed marked differences in the gut microbial composition between pancreatic cancer patients and healthy individuals, characterized by a significant reduction in short-chain fatty acid (SCFA)-producing bacteria and enrichment of inflammation-associated species. Furthermore, gut-derived microbes within pancreatic tumors are closely associated with immune microenvironment remodeling and gemcitabine resistance.

Similarly, gastric cancer patients exhibit distinct microbial profiles in both gastric fluid and tumor tissue compared with healthy controls-for instance, Helicobacter pylori enrichment-which may influence both tumorigenesis and neoadjuvant treatment efficacy. In colorectal cancer, Fusobacterium nucleatum and Peptostreptococcus anaerobius are significantly enriched in tumors resistant to immunotherapy, suggesting a key role of gut microbiota in treatment resistance. In hepatocellular carcinoma, intratumoral microbial subtypes are closely linked to tumor progression, and Klebsiella pneumoniae has been shown to promote hepatocarcinogenesis.

However, many key microbial species and their mechanistic roles in shaping the tumor microenvironment of digestive system cancers remain poorly understood, limiting the further clinical application of strategies such as neoadjuvant therapy in these patients. Therefore, a deeper investigation into the microbial characteristics of digestive system tumors and their correlation with neoadjuvant therapeutic response is of great clinical significance, particularly for identifying microbiome-based biomarkers that predict therapeutic efficacy and enable the selection of optimal candidate populations.

In summary, we have designed a prospective exploratory study to investigate the microbial characteristics and functional targets of digestive system cancers, aiming to develop and preliminarily validate a predictive model for identifying patient subgroups likely to benefit from neoadjuvant therapy. This study seeks to discover microbiome-associated biomarkers predictive of treatment efficacy and to expand the clinical application scope of neoadjuvant therapy in digestive system malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤80 years
* Pathologically confirmed diagnosis (via preoperative biopsy) of pancreatic cancer, gastric cancer, colorectal cancer, or esophageal cancer
* Imaging evaluation indicates borderline resectable or locally advanced disease, and the patient is scheduled to receive neoadjuvant therapy according to treatment guidelines
* Expected survival time > 3 months
* Hematologic function: neutrophil count > 1.5 × 10⁹/L
* Liver function:Total serum bilirubin ≤ 1.5 × upper limit of normal (ULN)；ALT and AST ≤ 2 × ULN
* Renal function: serum creatinine ≤ 1.5 × ULN
* No severe cardiovascular or cerebrovascular comorbidities and no psychiatric disorders

Exclusion Criteria:

* Physically unfit to undergo neoadjuvant chemotherapy
* Local recurrence or distant metastasis occurring within 1 month after surgery
* Impaired vital organ function, including but not limited to: Heart failure (NYHA Class III-IV); Myocardial infarction within the past 6 months; Severe arrhythmia; Respiratory failure
* Presence of another primary malignancy diagnosed within the past 5 years
* Pregnant or breastfeeding
* Inability to complete follow-up
* Active infection
* Severe constipation or sudden changes in bowel habits within the past 3 months
* Significant changes in dietary habits (e.g., meat-vegetable balance, meal timing, or frequency) within the past 3 months
* Medication history within the past 3 months including:Use of NSAIDs, immunosuppressants, antibiotics, traditional Chinese medicine, probiotics, or corticosteroids for ≥1 week; Use of proton pump inhibitors (PPIs) for more than 1 week within 1 month prior to sampling
* Refusal to sign the informed consent form

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pancreatic, gastric, or colorectal cancer who are scheduled to receive neoadjuvant therapy
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean fluorescence intensity of lipid raft staining in intratumoral immune cells measured by confocal immunofluorescence microscopy | 6 month
  Lipid raft staining intensity will be assessed by confocal immunofluorescence using cholera toxin subunit B (CTB). Quantification will be performed using ImageJ software and reported as mean fluorescence intensity per cell, averaged across representative fields per tumor sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Patients with esophageal, pancreatic, gastric, or colorectal cancer who are scheduled to receive neoadjuvant therapy, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided